CLINICAL TRIAL: NCT02869386
Title: Berlin PRehospital Or Usual Delivery of Acute Stroke Care - Functional Outcomes After Advanced Prehospital Stroke Care
Brief Title: Berlin PRehospital Or Usual Delivery of Acute Stroke Care
Acronym: B_PROUD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Center for Stroke Research Berlin (Other)
Responsible Party: Principal Investigator, Heinrich J Audebert, Prof. Dr. med., Charite University, Berlin, Germany
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B_PROUD
Record Dates: First submitted 2016-08-08; First posted 2016-08-16 (Estimated); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Stroke
Keywords: stroke; prehospital; telemedicine; thrombolysis; thrombectomy; endovascular treatment; functional outcome
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- STEMO deployment (Experimental): STEMO is a specialized stroke ambulance providing prehospital neurovascular expertise, a CT scanner, point-of-care testing, and telemedical support.
  Interventions: Procedure: STEMO
- Regular care (Active Comparator): Regular prehospital care consists of an ambulance. In suspected life-threatening cases an emergency physician is sent to the emergency scene in parallel.
  Interventions: Procedure: Regular care

INTERVENTIONS:
Procedure: STEMO — STEMO, the intervention, includes prehospital neurological emergency assessment with the option to perform CT and CT-angiography, start specialized treatment at the door-step of the patient's house, including thrombolysis with tissue Plasminogen Activator and blood pressure Management (choice of drug at discretion of treating physician), use telemedicine for further expertise as well as results of point-of-care laboratory, prenotification (e.g. for endovascular treatment), triage and transport.
  Arms: STEMO deployment
Procedure: Regular care — A regular ambulance, the comparator intervention, not equipped with advanced point-of-care laboratory or CT scanner, without telemedicine and not staffed with a neurologist.
  Arms: Regular care

SUMMARY:
Prehospital stroke care in specialized ambulances increases thrombolysis rates, reduces alarm-to-treatment times, and improves prehospital triage. Preliminary analyses suggest cost-effectiveness. However, scientific proof of improved functional outcome compared to usual care is still lacking. The objective of this trial is to show improved functional outcomes after deployment of the Stroke Emergency Mobile (STEMO) compared to regular care.

DETAILED DESCRIPTION:
This is a pragmatic, prospective, multi-center trial with blinded outcome assessment of treatment candidates three months after stroke. Treatment candidates will be defined as patients with final discharge diagnosis of cerebral ischemia, and onset-to-alarm time ≤4 hours, symptoms not resolved at time of ambulance arrival, and able to walk without assistance prior to emergency. These patients will be included if their emergency call from a predefined catchment area in Berlin, Germany, caused a stroke alarm at the dispatch center during STEMO hours (7am-11pm, Monday-Sunday). About 45% of STEMO dispatches will be handled by regular ambulances since STEMO will be already in operation creating the quasi-randomized control group.

B_PROUD uses data from the B-SPATIAL registry. The B-SPATIAL registry has started recruitment in January 2016. However, B_PROUD recruits patients with symptom onset October 1st, 2016 or later (because data access at the dispatch center had to be established first).

ELIGIBILITY:
Inclusion criteria:

1. Suspected acute stroke according to the dispatcher stroke identification algorithm during STEMO hours (7am-11pm, Monday-Sunday) and within the STEMO catchment area

   Inclusion criteria for primary study population:
2. Final diagnosis of ischemic stroke (ICD 10: I63) or TIA (ICD 10: G45 except G45.4)
3. Confirmed onset-to-alarm time ≤ 4 hours at dispatch
4. Pre-stroke modified Rankin scale ≤ 3 (being able to ambulate, in routine clinical care, patients with mRS up to 3 are usually deemed suitable for tissue plasminogen activator treatment)

Exclusion criteria:

1. Symptom remission until arrival of emergency medical service
2. Malignant or other severe primary disease with life expectancy < 1 year

   Exclusion criteria for primary study population:
3. Major surgery within 4 weeks before study inclusion
4. Confirmed stroke within 3 months before study inclusion
5. Absolute contraindications for thrombolysis AND thrombectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2019-10-24 (Actual); Study Completion 2019-10-24 (Actual)

PRIMARY OUTCOMES:
Modified Rankin Scale | 3 months
  Assessment of functional outcome over the entire range of the modified Rankin Scale
Co-primary 3-Month Outcome | 3 months
  The co-primary 3-month outcome includes the following range of outcomes:
  1. mRS 1-3 if available
  2. mRS 4-5 or (if mRS is missing) living in institution (information according registration office at 4 month after stroke)
  3. death.
  We will run a sensitivity analysis with the co-primary outcome and calculating all patients with missing mRS but still living under private address as mRS 1-3. The latter will help us to include information of patients still living at home but without mRS follow-up. All outcomes will be calculated with ordinal logistic regression.

SECONDARY OUTCOMES:
Thrombolysis rate | 3 months
Thrombectomy rate | 3 months
Diagnosis and treatment times (A) | 3 months
  Onset-to-treatment time
Diagnosis and treatment times (B) | 3 months
  onset-to-reperfusion time (for thrombectomy)
Diagnosis and treatment times (C) | 3 months
  alarm-to-imaging time
Diagnosis and treatment times (D) | 3 months
  alarm-to-treatment time
Diagnosis and treatment times (E) | 3 months
  imaging-to-treatment time
Cost-effectiveness (A) | 3 months
  Additional costs due to implementation and running of STEMO
Cost-effectiveness (B) | 3 months
  duration of hospital stay regarding acute treatment and rehabilitation
Cost-effectiveness (C) | 3 months
  hospital related costs
Cost-effectiveness (D) | 3 months
  costs of long-term care
Cost-effectiveness (E) | 3 months
  Additional costs due to implementation and running of STEMO, duration of hospital stay regarding acute treatment and rehabilitation, hospital related costs, costs of long-term care
Quality of life | Up to 5 years
  Assessment with European Quality of Life - 5 Dimensions (EQ-5D) in yearly intervals over 5 years to follow-up
Modified Rankin Scale shift analyses | 3 months
  Shift analyses for mRS ≤ 1 at 3 months in patients ≤ 80 years of age living at home without disability and mRS ≤ 2 at 3 months in patients > 80 years of age living at home with help or living in an institution
In-hospital mortality | 7 days
  Frequency of patients dying within the duration of the hospital stay after admission for stroke.
Death rate over time | 3 months
  Deaths over time will be determined and compared between groups using a Kaplan-Meier plot
Discharge status | 3 months
  Including in-hospital mortality among patients not included in the primary study population (patients with intracranial hemorrhages as well as patients receiving thrombolysis in stroke mimics)
Modified Rankin Scale in patients with intracranial hemorrhages | 3 months
  Assessment of functional outcome among patients with intracranial hemorrhages
Rate of emergency medical service deliveries to specialized facilities | 3 months
  Assessment for patients with acute ischemic stroke to hospitals with Stroke Unit, for patients with cerebral artery occlusion (internal carotid artery, M1 or proximal M2 segment of middle cerebral artery) to hospitals with thrombectomy facility, and for patients with intracerebral hemorrhage to hospitals with neurosurgery department.

OTHER OUTCOMES:
Symptomatic hemorrhage (A) | 3 months
  According to NINDS definition after 36 hours in patients receiving thrombolysis or thrombectomy
Symptomatic hemorrhage (B) | 3 months
  According to ECASS III definitions after 36 hours in patients receiving thrombolysis or thrombectomy

CONTACTS AND LOCATIONS:
Overall Officials: Heinrich Audebert, MD, Principal Investigator — Charité
Locations (1):
- Charite, Berlin, Germany

REFERENCES:
- [Background] Ebinger M, Winter B, Wendt M, Weber JE, Waldschmidt C, Rozanski M, Kunz A, Koch P, Kellner PA, Gierhake D, Villringer K, Fiebach JB, Grittner U, Hartmann A, Mackert BM, Endres M, Audebert HJ; STEMO Consortium. Effect of the use of ambulance-based thrombolysis on time to thrombolysis in acute ischemic stroke: a randomized clinical trial. JAMA. 2014 Apr 23-30;311(16):1622-31. doi: 10.1001/jama.2014.2850. PMID 24756512
- [Background] Krebes S, Ebinger M, Baumann AM, Kellner PA, Rozanski M, Doepp F, Sobesky J, Gensecke T, Leidel BA, Malzahn U, Wellwood I, Heuschmann PU, Audebert HJ. Development and validation of a dispatcher identification algorithm for stroke emergencies. Stroke. 2012 Mar;43(3):776-81. doi: 10.1161/STROKEAHA.111.634980. Epub 2012 Jan 5. PMID 22223240
- [Background] Ebinger M, Fiebach JB, Audebert HJ. Mobile computed tomography: prehospital diagnosis and treatment of stroke. Curr Opin Neurol. 2015 Feb;28(1):4-9. doi: 10.1097/WCO.0000000000000165. PMID 25490196
- [Background] Wendt M, Ebinger M, Kunz A, Rozanski M, Waldschmidt C, Weber JE, Winter B, Koch PM, Freitag E, Reich J, Schremmer D, Audebert HJ; STEMO Consortium. Improved prehospital triage of patients with stroke in a specialized stroke ambulance: results of the pre-hospital acute neurological therapy and optimization of medical care in stroke study. Stroke. 2015 Mar;46(3):740-5. doi: 10.1161/STROKEAHA.114.008159. Epub 2015 Jan 29. PMID 25634000
- [Background] Kunz A, Ebinger M, Geisler F, Rozanski M, Waldschmidt C, Weber JE, Wendt M, Winter B, Zieschang K, Fiebach JB, Villringer K, Erdur H, Scheitz JF, Tutuncu S, Bollweg K, Grittner U, Kaczmarek S, Endres M, Nolte CH, Audebert HJ. Functional outcomes of pre-hospital thrombolysis in a mobile stroke treatment unit compared with conventional care: an observational registry study. Lancet Neurol. 2016 Sep;15(10):1035-43. doi: 10.1016/S1474-4422(16)30129-6. Epub 2016 Jul 16. PMID 27430529
- [Background] Ebinger M, Harmel P, Nolte CH, Grittner U, Siegerink B, Audebert HJ. Berlin prehospital or usual delivery of acute stroke care - Study protocol. Int J Stroke. 2017 Aug;12(6):653-658. doi: 10.1177/1747493017700152. Epub 2017 Mar 22. PMID 28649936
- [Background] Kunz A, Nolte CH, Erdur H, Fiebach JB, Geisler F, Rozanski M, Scheitz JF, Villringer K, Waldschmidt C, Weber JE, Wendt M, Winter B, Zieschang K, Grittner U, Kaczmarek S, Endres M, Ebinger M, Audebert HJ. Effects of Ultraearly Intravenous Thrombolysis on Outcomes in Ischemic Stroke: The STEMO (Stroke Emergency Mobile) Group. Circulation. 2017 May 2;135(18):1765-1767. doi: 10.1161/CIRCULATIONAHA.117.027693. No abstract available. PMID 28461420
- [Derived] Piccininni M, Kurth T, Audebert HJ, Rohmann JL. The Effect of Mobile Stroke Unit Care on Functional Outcomes: An Application of the Front-door Formula. Epidemiology. 2023 Sep 1;34(5):712-720. doi: 10.1097/EDE.0000000000001642. Epub 2023 Jun 30. PMID 37462471
- See also: Prehospital Thrombolysis: A Manual from Berlin (2013) — http://www.jove.com/video/50534/prehospital-thrombolysis-a-manual-from-berlin